CLINICAL TRIAL: NCT03619057
Title: Voice Tessitura and Size of the Required Laryngeal Mask
Acronym: EVG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: EVG
Record Dates: First submitted 2018-07-30; First posted 2018-08-07 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Laryngeal Masks
MeSH Terms: interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- > 18 years
  Interventions: Other: General anesthesia with laryngeal mask i-gel
- 10 to 18 years
  Interventions: Other: General anesthesia with laryngeal mask i-gel

INTERVENTIONS:
Other: General anesthesia with laryngeal mask i-gel — General anesthesia with laryngeal mask i-gel

SUMMARY:
The choice of the size of the laryngeal mask (i-gel) is based on the weight. Even following the weight recommendations, it is quite common to choose a mask that is too big or too small, which leads to ventilation leaks (too small), or insertion failures (too big) and leads to a change of mask for bigger or smaller.

The i-gel are laryngeal masks (2nd generation) which consist of gel and have been designed by molding on larynx corpses. The masks are not inflatable (so not adaptable).

I-gel masks are used in adult and pediatric patients for weights ranging from 2 Kg to over 90 Kg to provide ventilation during general anesthesia.

Patients with a deep voice probably need a larger laryngeal mask than their weight alone suggests.

The investigators propose to measure the lowest sound emitted by the patient because it would seem logical that the larger the larynx is, the more the voice is serious.

This hypothesis will be verified a posteriori by the size of the laryngeal mask used and adapted by comparing it to the range of the voice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 10 years
* Planned surgical procedure with the use of a laryngeal mask

Exclusion Criteria:

• Refusal to participate in the study.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients up to 10 years old with planned surgery and anticipated use of laryngeal mask i-gel.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-24 (Actual)

PRIMARY OUTCOMES:
Concordance between the weight and the tessitura threshold | 1 day
  Concordance between the size of the mask proposed as a function of the weight and that determined after determination of the tessitura threshold for each mask size by ROC curves.

SECONDARY OUTCOMES:
Determining the tessitura threshold corresponding to each mask size | 1 day
  tessitura threshold (the most serious sound emitted by the patient) corresponding to each mask size

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Villeneuve-Saint-Georges, Villeneuve-Saint-Georges, France

IPD SHARING:
Plan to Share IPD: No